CLINICAL TRIAL: NCT02876328
Title: Partnership for Research on Ebola VACcinations (PREVAC)
Brief Title: Partnership for Research on Ebola VACcinations
Acronym: PREVAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Partnership for Research on Ebola Virus in Liberia (PREVAIL) (Network); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); London School of Hygiene and Tropical Medicine (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C15-33; PREVACEBL3005 (Other: LSHTM)
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Ebola Virus Disease
Keywords: Ebola Vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ad26.ZEBOV (rHAd26) vaccine + MVA-BN-Filo (MVA) boost (Experimental): Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Placebo (0.5 mL) (Placebo Comparator): Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Interventions: Biological: Placebo
- rVSVΔG-ZEBOV-GP (rVSV) vaccine + placebo boost (Experimental): Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by a placebo boost at Day 56.
  Interventions: Biological: rVSVΔG-ZEBOV-GP; Biological: Placebo
- rVSVΔG-ZEBOV-GP (rVSV) vaccine + rVSV boost (Experimental): Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by an rVSV boost at Day 56.
  Interventions: Biological: rVSVΔG-ZEBOV-GP; Biological: rVSV boost
- Placebo (1 mL) (Placebo Comparator): Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV — 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm for adults or the thigh for children
  Other Names: rHAd26
  Arms: Ad26.ZEBOV (rHAd26) vaccine + MVA-BN-Filo (MVA) boost
Biological: MVA-BN-Filo — 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm for adults or the thigh for children
  Other Names: MVA; MVA-mBN226B
  Arms: Ad26.ZEBOV (rHAd26) vaccine + MVA-BN-Filo (MVA) boost
Biological: rVSVΔG-ZEBOV-GP — 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm for adults or the thigh for children
  Other Names: rVSV; V920
  Arms: rVSVΔG-ZEBOV-GP (rVSV) vaccine + placebo boost; rVSVΔG-ZEBOV-GP (rVSV) vaccine + rVSV boost
Biological: Placebo — 0.5 mL or 1 mL (depending upon the arm) sterile normal saline administered by intramuscular (IM) injection into the upper arm for adults or the thigh for children
  Arms: Placebo (0.5 mL); Placebo (1 mL); rVSVΔG-ZEBOV-GP (rVSV) vaccine + placebo boost
Biological: rVSV boost — 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm for adults or the thigh for children
  Other Names: rVSVΔG-ZEBOV-GP; rVSV; V920
  Arms: rVSVΔG-ZEBOV-GP (rVSV) vaccine + rVSV boost

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of three vaccine strategies that may prevent Ebola virus disease (EVD) events in children and adults. Participants will receive either the Ad26.ZEBOV (rHAd26) vaccine with a MVA-BN-Filo (MVA) boost, or the rVSVΔG-ZEBOV-GP (rVSV) vaccine with or without boosting, or placebo.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and immunogenicity of two Ebola virus disease (EVD) vaccines, Ad26.ZEBOV (rHAd26) and rVSVΔG-ZEBOV-GP (rVSV), in children and adults. These vaccines will be studied using three different strategies: the rHAd26 vaccine plus a MVA-BN-Filo (MVA) boost, and the rVSV vaccine with or without boosting.

Participants will be randomized into five groups: the Ad26.ZEBOV vaccine with an MVA boost, the rVSV vaccine with or without boosting, or one of two placebo groups. At Day 0 (study entry), participants will receive the Ad26.ZEBOV vaccine, the rVSV vaccine, or placebo.

At Day 56, participants assigned to the rVSV vaccine without a boost and the two placebo groups will receive placebo. Those initially given the Ad26.ZEBOV vaccine will receive the MVA boost. Those assigned to the boosted rVSV group will receive the rVSV boost.

Additional study visits will occur on Days 7, 14, 28, and 63, and at Months 3, 6, 12, 24, 36, 48, and 60. Study visits may include blood collection and other assessments.

Some participants may take part in substudies, which will include blood or saliva collection.

After the Month 12 visit, during the long-term follow-up, the participants who received the placebo will be vaccinated with a single dose of rVSVΔG-ZEBOV-GP vaccine in Liberia and Mali and with the Ad26.ZEBOV/MVA-BN-Filo vaccine strategy in Guinea and Sierra Leone. The participants who received an incomplete Ad26.ZEBOV/MVA-BN-Filo vaccine strategy will be offered a single dose of the Ad26.ZEBOV or MVA-BN-Filo vaccine in Guinea and Sierra Leone and a single dose of rVSVΔG-ZEBOV-GP in Liberia and Mali.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent
* Age greater than or equal to 1 year
* Planned residency in the area of the study site for the next 12 months
* Willingness to comply with the protocol requirements

Exclusion Criteria:

* Fever greater than 38º Celsius
* History of EVD (self-report)
* Pregnancy (a negative urine pregnancy test is required for females of child-bearing potential, i.e., females who have experienced menarche or who are aged 14 years and older)
* Positive HIV test for participants less than 18 years of age
* Reported current breast-feeding
* Prior vaccination against Ebola (self-report)
* Any vaccination in the past 28 days or planned within the 28 days after randomization (initial vaccination)
* In the judgement of the clinician, any clinically significant acute/chronic condition that would limit the ability of the participant to meet the requirements of the study protocol

Inclusion Criteria for Revaccination Post 12 Month Visit:

* Participants who received the placebo
* Participants who received an incomplete Ad26.ZEBOV/MVA-BN-Filo vaccine strategy

Temporary Exclusion Criteria for Revaccination Post 12 Month Visit:

* Fever greater than 38º Celsius
* Pregnancy (a negative urine pregnancy test is required for females of child-bearing potential, i.e., females who have experienced menarche or who are aged 14 years and older)
* Reported current breast-feeding (self-report)
* Any vaccination in the past 28 days or planned within the 28 days after trial vaccination

Exclusion Criteria for Revaccination Post 12 Month Visit:

* EVD notified in the electronic case report form
* For minor participants: change in HIV status since enrollment (self-report)
* Previous Ebola vaccination outside of the study including incomplete vaccine strategies
* Known medical history or significant risk factors for a thrombotic and/or thrombocytopenic event (for participants who will receive the Ad26.ZEBOV or MVA-BN-Filo vaccine)

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4789 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yazdan Yazdanpannah, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Abdoul Habib Beavogui, Principal Investigator — Centre de Formation et de Recherche en Santé Rurale de Mafèrinyah; Mark Kieh, Principal Investigator — Redemption Hospital; Bailah Leigh, Principal Investigator — University of Sierra Leone; Stephen B. Kennedy, Principal Investigator — Redemption Hospital; Seydou Doumbia, Principal Investigator — Universite des Sciences, des Techniques et des Technologies de Bamako; Samba O. Sow, Principal Investigator — Centre pour le Developpement des Vaccins
Locations (6):
- Guinea (2):
  - Centre national de formation et de recherche en santé rurale (Maferyniah), Conakry
  - Landreah, Conakry
- The Redemption Hospital, Monrovia, Liberia
- Mali (2):
  - Centre pour le Développement des Vaccins (CVD), Bamako
  - University Clinical Research Center (UCRC), Bamako
- Mambolo Clinic, Kapesseh, Sierra Leone

REFERENCES:
- [Result] Badio M, Lhomme E, Kieh M, Beavogui AH, Kennedy SB, Doumbia S, Leigh B, Sow SO, Diallo A, Fusco D, Kirchoff M, Termote M, Vatrinet R, Wentworth D, Esperou H, Lane HC, Pierson J, Watson-Jones D, Roy C, D'Ortenzio E, Greenwood B, Chene G, Richert L, Neaton JD, Yazdanpanah Y; PREVAC study team. Partnership for Research on Ebola VACcination (PREVAC): protocol of a randomized, double-blind, placebo-controlled phase 2 clinical trial evaluating three vaccine strategies against Ebola in healthy volunteers in four West African countries. Trials. 2021 Jan 23;22(1):86. doi: 10.1186/s13063-021-05035-9. PMID 33485369
- [Result] PREVAC Study Team; Kieh M, Richert L, Beavogui AH, Grund B, Leigh B, D'Ortenzio E, Doumbia S, Lhomme E, Sow S, Vatrinet R, Roy C, Kennedy SB, Faye S, Lees S, Millimouno NP, Camara AM, Samai M, Deen GF, Doumbia M, Esperou H, Pierson J, Watson-Jones D, Diallo A, Wentworth D, McLean C, Simon J, Wiedemann A, Dighero-Kemp B, Hensley L, Lane HC, Levy Y, Piot P, Greenwood B, Chene G, Neaton J, Yazdanpanah Y. Randomized Trial of Vaccines for Zaire Ebola Virus Disease. N Engl J Med. 2022 Dec 29;387(26):2411-2424. doi: 10.1056/NEJMoa2200072. Epub 2022 Dec 14. PMID 36516078
- [Derived] Kpetigo AD, Alexandre M, Camara A, Beavogui A, Doumbia S, Kieh M, Leigh B, Sow S, Wittkop L, Soutthiphong AA, Berry IM, Fleck S, Akoo P, Hamze B, Watson-Jones D, Kuhn JH, Greenwood B, Richert L, Yazdanpanah Y, Levy Y, Thiebaut R, Prague M; PREVAC Study Team; Lhomme E. Effect of the time of day for vaccination on the immune response to Ebola Virus Disease vaccines: A modeling study from PREVAC randomized trial. PLoS Negl Trop Dis. 2026 Jan 30;20(1):e0013950. doi: 10.1371/journal.pntd.0013950. Online ahead of print. PMID 41616038
- [Derived] Valayer S, Alexandre M, Prague M, Beavogui AH, Doumbia S, Kieh M, Greenwood B, Leigh B, Poupelin M, Schwimmer C, Sow SO, Berry IM, Kuhn JH, Fusco D, Cauwelaert ND, Watson-Jones D, Thiebaut R, Levy Y, Yazdanpanah Y, Richert L, Lhomme E; PREVAC study team. Evaluation of waning of IgG antibody responses after rVSVDeltaG-ZEBOV-GP and Ad26.ZEBOV, MVA-BN-Filo Ebola virus disease vaccines: a modelling study from the PREVAC randomized trial. Emerg Microbes Infect. 2025 Dec;14(1):0. doi: 10.1080/22221751.2024.2432353. Epub 2024 Dec 9. PMID 39559990
- [Derived] Wiedemann A, Lhomme E, Huchon M, Foucat E, Bererd-Camara M, Guillaumat L, Yaradouno M, Tambalou J, Rodrigues C, Ribeiro A, Beavogui AH, Lacabaratz C, Thiebaut R, Richert L, Levy Y; Prevac study team. Long-term cellular immunity of vaccines for Zaire Ebola Virus Diseases. Nat Commun. 2024 Sep 3;15(1):7666. doi: 10.1038/s41467-024-51453-z. PMID 39227399
- [Derived] Lee AW, Liu K, Lhomme E, Blie J, McCullough J, Onorato MT, Connor L, Simon JK, Dubey S, VanRheenen S, Deutsch J, Owens A, Morgan A, Welebob C, Hyatt D, Nair S, Hamze B, Guindo O, Sow SO, Beavogui AH, Leigh B, Samai M, Akoo P, Serry-Bangura A, Fleck S, Secka F, Lowe B, Watson-Jones D, Roy C, Hensley LE, Kieh M, Coller BG; PREVAC Study Team. Immunogenicity and Vaccine Shedding After 1 or 2 Doses of rVSVDeltaG-ZEBOV-GP Ebola Vaccine (ERVEBO(R)): Results From a Phase 2, Randomized, Placebo-controlled Trial in Children and Adults. Clin Infect Dis. 2024 Apr 10;78(4):870-879. doi: 10.1093/cid/ciad693. PMID 37967326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were enrolled at 6 sites in 4 countries: Guinea at 2 sites (Landreah and Maferinyah), Liberia (Redemption Hospital), Mali at 2 sites (Center for Vaccine Development and the University Clinical Research Center), and Sierra Leone (Mambolo). Total enrollment includes participants enrolled in all versions of the protocol, but only participants enrolled in version 4.0 of the protocol are included in the primary outcome analysis.
Pre-assignment Details: 4789 participants were enrolled in the study, however, only 4786 participants are part of the data analysis.
Groups:
- Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v4.0): Protocol Version 4.0
  Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Ad26.ZEBOV: 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm
  MVA-BN-Filo: 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm
- Placebo (0.5 mL) - Adults (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Adults (v4.0): Protocol Version 4.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by a placebo boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Adults (v4.0): Protocol Version 4.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by an rVSV boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm
  rVSV boost: 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm
- Placebo (1 mL) - Adults (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v4.0): Protocol Version 4.0
  Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Ad26.ZEBOV: 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm or the thigh
  MVA-BN-Filo: 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm or the thigh
- Title: Placebo (0.5 mL) - Children (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or the thigh
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Children (v4.0): Protocol Version 4.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by a placebo boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm or the thigh
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or the thigh
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Children (v4.0): Protocol Version 4.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by an rVSV boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm or the thigh
  rVSV boost: 1 mL at a nominal dose of 2x10^7 pfu/mL administered by intramuscular (IM) injection into the upper arm or the thigh
- Placebo (1 mL) - Children (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or the thigh
- Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v3.0): Protocol Version 3.0
  Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Ad26.ZEBOV: 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm
  MVA-BN-Filo: 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm
- Placebo (0.5 mL) - Adults (v3.0): Protocol Version 3.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Adults (v3.0): Protocol Version 3.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by a placebo boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Adults (v3.0): Protocol Version 3.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by an rVSV boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm
  rVSV boost: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm
- Placebo (1 mL) - Adults (v3.0): Protocol Version 3.0 Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v3.0): Protocol Version 3.0
  Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Ad26.ZEBOV: 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm or thigh
  MVA-BN-Filo: 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm or thigh
- Placebo (0.5 mL) - Children (v3.0): Protocol Version 3.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or thigh
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0): Protocol Version 3.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by a placebo boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm or thigh
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Children (v3.0): Protocol Version 3.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by an rVSV boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm or thigh
  rVSV boost: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm or thigh
- Placebo (1 mL) - Children (v3.0): Protocol Version 3.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or thigh
- Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v2.0): Protocol Version 2.0
  Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Ad26.ZEBOV: 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm
  MVA-BN-Filo: 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm
- Placebo (0.5 mL) - Adults (v2.0): Protocol Version 2.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v2.0): Protocol Version 2.0
  Participants will receive the Ad26.ZEBOV (rHAd26) vaccine at Day 0 followed by an MVA-BN-Filo (MVA) boost at Day 56.
  Ad26.ZEBOV: 0.5 mL at a dose of 5x10^10 vp administered by intramuscular (IM) injection into the upper arm or thigh
  MVA-BN-Filo: 0.5 mL at a dose of 1x10^8 InfU administered by intramuscular (IM) injection into the upper arm or thigh
- Placebo (0.5 mL) - Children (v2.0): Protocol Version 2.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or thigh
Period: Overall Study
Arm/Group | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v4.0) | Placebo (0.5 mL) - Adults (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Adults (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Adults (v4.0) | Placebo (1 mL) - Adults (v4.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v4.0) | Title: Placebo (0.5 mL) - Children (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Children (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Children (v4.0) | Placebo (1 mL) - Children (v4.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v3.0) | Placebo (0.5 mL) - Adults (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Adults (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Adults (v3.0) | Placebo (1 mL) - Adults (v3.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v3.0) | Placebo (0.5 mL) - Children (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Children (v3.0) | Placebo (1 mL) - Children (v3.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v2.0) | Placebo (0.5 mL) - Adults (v2.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v2.0) | Placebo (0.5 mL) - Children (v2.0)
Started | 396 | 221 | 395 | 197 | 191 | 403 | 179 | 407 | 202 | 210 | 187 | 99 | 177 | 99 | 100 | 227 | 107 | 237 | 108 | 107 | 324 | 172 | 34 | 7
Completed (For the primary outcome, Completed is defined as attending the 12 month visit.) | 379 | 208 | 378 | 188 | 181 | 388 | 175 | 395 | 192 | 202 | 182 | 98 | 172 | 95 | 96 | 223 | 102 | 227 | 106 | 105 | 312 | 164 | 33 | 7
Not Completed | 17 | 13 | 17 | 9 | 10 | 15 | 4 | 12 | 10 | 8 | 5 | 1 | 5 | 4 | 4 | 4 | 5 | 10 | 2 | 2 | 12 | 8 | 1 | 0
Not completed — Death | 2 | 1 | 3 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 3 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Missed 12 Month Visit | 15 | 10 | 11 | 6 | 10 | 14 | 3 | 8 | 9 | 5 | 4 | 1 | 5 | 4 | 4 | 4 | 3 | 6 | 2 | 2 | 11 | 7 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (0.5 mL) - Children (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or the thigh
- Placebo (1 mL) - Children (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0): Protocol Version 3.0
  Participants will receive the rVSVΔG-ZEBOV-GP (rVSV) vaccine at Day 0 followed by a placebo boost at Day 56.
  rVSVΔG-ZEBOV-GP: 1 mL of a 1:2 diluted 2x10^7 pfu/mL nominal dose administered by intramuscular (IM) injection into the upper arm or thigh
  Placebo: 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or thigh
- Total: Total of all reporting groups
Arm/Group | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v4.0) | Placebo (0.5 mL) - Adults (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Adults (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Adults (v4.0) | Placebo (1 mL) - Adults (v4.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v4.0) | Placebo (0.5 mL) - Children (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Children (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Children (v4.0) | Placebo (1 mL) - Children (v4.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v3.0) | Placebo (0.5 mL) - Adults (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Adults (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Adults (v3.0) | Placebo (1 mL) - Adults (v3.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v3.0) | Placebo (0.5 mL) - Children (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Children (v3.0) | Placebo (1 mL) - Children (v3.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v2.0) | Placebo (0.5 mL) - Adults (v2.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v2.0) | Placebo (0.5 mL) - Children (v2.0) | Total
Number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 403 | 179 | 407 | 202 | 210 | 187 | 99 | 177 | 99 | 100 | 227 | 107 | 237 | 108 | 107 | 324 | 172 | 34 | 7 | 4786
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Adults and children are analyzed separately.
  years
    Adults: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Adults | 27 [21 to 40] | 28 [20 to 38] | 27 [20 to 39] | 26 [20 to 35] | 26 [21 to 38] |  |  |  |  |  | 30 [23 to 44] | 31 [23 to 40] | 29 [22 to 39] | 28 [22 to 43] | 28 [22 to 39] |  |  |  |  |  | 27 [22 to 37] | 27 [22 to 37] |  |  | 27 [21 to 39]
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Children |  |  |  |  |  | 8 [4 to 13] | 8 [4 to 13] | 9 [4 to 12] | 8 [3 to 13] | 8 [4 to 13] |  |  |  |  |  | 12 [8 to 15] | 12 [8 to 15] | 12 [8 to 15] | 12 [7 to 15] | 12 [7 to 14] |  |  | 14 [13 to 16] | 14 [12 to 15] | 10 [5 to 14]
Age, Customized [Count of Participants; unit: Participants]
  1-4 years | 0 | 0 | 0 | 0 | 0 | 137 | 59 | 123 | 71 | 77 | 0 | 0 | 0 | 0 | 0 | 25 | 12 | 24 | 9 | 12 | 0 | 0 | 0 | 0 | 549
  5-11 years | 0 | 0 | 0 | 0 | 0 | 127 | 59 | 146 | 65 | 70 | 0 | 0 | 0 | 0 | 0 | 76 | 37 | 86 | 43 | 41 | 0 | 0 | 0 | 0 | 750
  12-17 years | 0 | 0 | 0 | 0 | 0 | 139 | 61 | 138 | 66 | 63 | 0 | 0 | 0 | 0 | 0 | 126 | 58 | 127 | 56 | 54 | 0 | 0 | 34 | 7 | 929
  Adults >18 years | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Adults and children are analyzed separately.
  Participants
    Adults: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Adults: Female | 171 | 106 | 182 | 87 | 81 |  |  |  |  |  | 99 | 45 | 75 | 43 | 49 |  |  |  |  |  | 120 | 60 |  |  | 1118
    Adults: Male | 225 | 115 | 213 | 110 | 110 |  |  |  |  |  | 88 | 54 | 102 | 56 | 51 |  |  |  |  |  | 204 | 112 |  |  | 1440
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Children: Female |  |  |  |  |  | 186 | 87 | 185 | 85 | 95 |  |  |  |  |  | 122 | 48 | 117 | 55 | 53 |  |  | 19 | 5 | 1057
    Children: Male |  |  |  |  |  | 217 | 92 | 222 | 117 | 115 |  |  |  |  |  | 105 | 59 | 120 | 53 | 54 |  |  | 15 | 2 | 1171
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: Adults and children are analyzed separately.
  Participants
    Guinea: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Guinea | 121 | 72 | 130 | 66 | 63 |  |  |  |  |  | 144 | 80 | 141 | 77 | 76 |  |  |  |  |  | 158 | 84 |  |  | 1212
    Liberia: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Liberia | 73 | 43 | 70 | 35 | 38 |  |  |  |  |  | 43 | 19 | 36 | 22 | 24 |  |  |  |  |  | 166 | 88 |  |  | 657
    Mali: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Mali | 81 | 48 | 84 | 41 | 38 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  | 0 | 0 |  |  | 292
    Sierra Leone: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Sierra Leone | 121 | 58 | 111 | 55 | 52 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  | 0 | 0 |  |  | 397
Region of Enrollment [Count of Participants; unit: Participants] — Population: Adults and children are analyzed separately.
  Participants
    Guinea: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Guinea |  |  |  |  |  | 163 | 71 | 156 | 77 | 79 |  |  |  |  |  | 160 | 72 | 163 | 76 | 77 |  |  | 17 | 4 | 1115
    Liberia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Liberia |  |  |  |  |  | 64 | 25 | 66 | 33 | 30 |  |  |  |  |  | 67 | 35 | 74 | 32 | 30 |  |  | 17 | 3 | 476
    Mali: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Mali |  |  |  |  |  | 95 | 40 | 94 | 46 | 51 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 326
    Sierra Leone: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Sierra Leone |  |  |  |  |  | 81 | 43 | 91 | 46 | 50 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 311
HIV Positive [Count of Participants; unit: Participants] — Population: Adults and children are analyzed separately. HIV positive minors were not included in the study.
  Participants
    Adults: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 187 | 99 | 177 | 99 | 100 | 0 | 0 | 0 | 0 | 0 | 324 | 172 | 0 | 0 | 2558
    Adults | 6 | 1 | 13 | 2 | 3 |  |  |  |  |  | 5 | 2 | 4 | 2 | 2 |  |  |  |  |  | 6 | 8 |  |  | 54
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 227 | 107 | 237 | 108 | 107 | 0 | 0 | 34 | 7 | 2228
    Children |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0
Number of Participants with Results for Ebola IgG Concentration (Version 4) [Count of Participants; unit: Participants] — Population: The number of participants analyzed reflects the number of participants with baseline Ebola IgG results from Version 4.0 of the protocol. Adults and children were analyzed separately.
  Participants
    Adults: number analyzed (Participants) | 396 | 221 | 395 | 197 | 191 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1400
    Adults | 394 | 220 | 388 | 197 | 189 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1388
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 403 | 179 | 407 | 202 | 210 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1401
    Children |  |  |  |  |  | 398 | 177 | 401 | 200 | 209 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1385
Number of Participants with Ebola IgG Concentration < 66.96 EU/mL (Version 4) [Count of Participants; unit: Participants] — 66.96 EU/mL is the lower limit of quantification for the Filovirus Animal Nonclinical Group (FANG) enzyme-linked immunosorbent assay (ELISA) Population: The number of participants analyzed reflects the number of participants with baseline Ebola IgG results from Version 4.0 of the protocol. Adults and children were analyzed separately.
  Participants
    Adults: number analyzed (Participants) | 394 | 220 | 388 | 197 | 189 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1388
    Adults | 142 | 78 | 144 | 66 | 68 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 498
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 398 | 177 | 401 | 200 | 209 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1385
    Children |  |  |  |  |  | 198 | 87 | 187 | 97 | 101 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 670
Number of Participants with Ebola IgG Concentration >= 200 EU/mL (Version 4.0) [Count of Participants; unit: Participants] — Population: The number of participants analyzed reflects the number of participants with baseline Ebola IgG results from Version 4.0 of the protocol. Adults and children were analyzed separately.
  Participants
    Adults: number analyzed (Participants) | 394 | 220 | 388 | 197 | 189 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1388
    Adults | 50 | 38 | 58 | 32 | 30 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 208
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 398 | 177 | 401 | 200 | 209 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1385
    Children |  |  |  |  |  | 43 | 22 | 47 | 19 | 32 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 163
Median Ebola IgG Concentration (Version 4.0) [Median (Inter-Quartile Range); unit: EU/mL] — Population: The number of participants analyzed reflects the number of participants with baseline Ebola IgG results from Version 4.0 of the protocol. Adults and children were analyzed separately.
  EU/mL
    Adults: number analyzed (Participants) | 394 | 220 | 388 | 197 | 189 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1388
    Adults | 94 [43 to 149] | 99 [49 to 158] | 92 [45 to 145] | 94 [46 to 143] | 94 [47 to 149] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 95 [46 to 148]
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 398 | 177 | 401 | 200 | 209 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1385
    Children |  |  |  |  |  | 67 [29 to 127] | 68 [33 to 114] | 74 [33 to 122] | 69 [33 to 122] | 78 [33 to 151] |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 70 [32 to 128]
Geometric Mean Ebola IgG Concentration (Version 4.0) [Geometric Mean (Standard Deviation); unit: EU/mL] — Population: The number of participants analyzed reflects the number of participants with baseline Ebola IgG results from Version 4.0 of the protocol. Adults and children were analyzed separately.
  EU/mL
    Adults: number analyzed (Participants) | 394 | 220 | 388 | 197 | 189 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1388
    Adults | 85 (2.7) | 92 (2.8) | 87 (2.7) | 91 (2.7) | 87 (2.8) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 88 (2.7)
    Children: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 398 | 177 | 401 | 200 | 209 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1385
    Children |  |  |  |  |  | 63 (3.0) | 66 (2.8) | 67 (3.0) | 67 (3.1) | 73 (3.1) |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 66 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ebola Virus Glycoprotein (GP-EBOV) Antibody Response
Description: Antibody responder at 12 months is defined as a participant who experiences a 4-fold increase in antibody level from baseline and for whom the antibody level at 12 months is greater than or equal to 200 EU/mL.
Time Frame: Measured through Month 12
Population: The analysis population only includes participants from version 4.0 of the protocol. Adults and children are analyzed separately.
  Participants with a missing baseline or 12-month antibody result are excluded. Participants with elevated antibody levels at baseline were not excluded. The placebo group is pooled. Percentages of participants that do not yield whole numbers are the result of rounding.
Measure: Number; unit: percentage of participants
Groups:
- Protocol Version 4.0 Ad26/MVA: Ad26.ZEBOV first dose (0.5 mL) followed by an MVA-BN-Filo second dose (0.5 mL) at 56 days
- Protocol Version 4.0 rVSV: rVSVΔG-ZEBOV-GP first dose (1 mL) followed by placebo second dose (1 mL) at 56 days
- Protocol Version 4.0 rVSV Boost: rVSVΔG-ZEBOV-GP first dose(1 mL) followed by an rVSVΔG-ZEBOV-GP dose (1 mL) at 56 days
- Protocol Version 4.0 Pooled Placebo: Placebo dose (0.5 mL or 1 mL) followed by a placebo second dose (0.5 mL or 1 mL) at 56 days
Arm/Group | Protocol Version 4.0 Ad26/MVA | Protocol Version 4.0 rVSV | Protocol Version 4.0 rVSV Boost | Protocol Version 4.0 Pooled Placebo
Number analyzed (Participants) | 755 | 756 | 374 | 741
percentage of participants
  Adults: number analyzed (Participants) | 374 | 371 | 185 | 377
  Adults | 40.9 | 75.7 | 81.1 | 2.7
  Children: number analyzed (Participants) | 381 | 385 | 189 | 364
  Children | 78.5 | 87.3 | 92.6 | 3.6
Statistical Analysis 1: Comparison: Protocol Version 4.0 Ad26/MVA vs Protocol Version 4.0 rVSV vs Protocol Version 4.0 rVSV Boost vs Protocol Version 4.0 Pooled Placebo; Analysis applies to both adults and children; Test type: Superiority; p < .001, Cochran-Mantel-Haenszel — Each active group is compared to placebo using a 2-sided .0167 significance level; Analyses are stratified by site

2. Secondary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: SAEs as defined in the protocol
Time Frame: Measured through Month 60
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With Ebola Virus Glycoprotein (GP-EBOV) Antibody Response
Description: Antibodies to the Ebola virus glycoprotein will be measured with the Filovirus Animal Nonclinical Group (FANG) ELISA assay if available. Other assays may also be used.
Time Frame: Measured through Month 60
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months for the Primary Outcome. Adverse events will be collected through the end of the study (60 months). A full summary will be provided when the study is complete.
Description: AEs of grade 1 or 2 severity other than injection site reactions and targeted symptoms were not collected.
  Systematically assessed AEs were collected via standard checklist.
Groups:
- Pooled Placebo (0.5 mL or 1 mL) - Adults (v4.0); Pooled Placebo (0.5 mL or 1 mL) - Children (v4.0): Protocol Version 4.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL or 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- Pooled Placebo (0.5 mL or 1 mL) - Adults (v3.0): Protocol Version 3.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL or 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm
- Pooled Placebo (0.5 mL or 1 mL) - Children (v3.0): Protocol Version 3.0
  Participants will receive placebo at Day 0 followed by a placebo boost at Day 56.
  Placebo: 0.5 mL or 1 mL sterile normal saline administered by intramuscular (IM) injection into the upper arm or thigh
Arm/Group | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v4.0) | Pooled Placebo (0.5 mL or 1 mL) - Adults (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Adults (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Adults (v4.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v4.0) | Pooled Placebo (0.5 mL or 1 mL) - Children (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Children (v4.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Children (v4.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v3.0) | Pooled Placebo (0.5 mL or 1 mL) - Adults (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Adults (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Adults (v3.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v3.0) | Pooled Placebo (0.5 mL or 1 mL) - Children (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Children (v3.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v2.0) | Placebo (0.5 mL) - Adults (v2.0) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v2.0) | Placebo (0.5 mL) - Children (v2.0)
All-Cause Mortality (participants affected / at risk) | 2/396 | 1/412 | 3/395 | 0/197 | 0/403 | 2/389 | 3/407 | 0/202 | 1/187 | 0/199 | 0/177 | 0/99 | 0/227 | 1/214 | 1/237 | 0/108 | 0/324 | 1/172 | 0/34 | 0/7
Serious Adverse Events (participants affected / at risk) | 14/396 | 5/412 | 6/395 | 1/197 | 5/403 | 8/389 | 9/407 | 3/202 | 12/187 | 6/199 | 6/177 | 2/99 | 4/227 | 7/214 | 6/237 | 1/108 | 6/324 | 5/172 | 1/34 | 0/7
Other Adverse Events (participants affected / at risk) | 296/396 | 291/412 | 320/395 | 155/197 | 341/403 | 298/389 | 350/407 | 179/202 | 142/187 | 151/199 | 148/177 | 80/99 | 167/227 | 143/214 | 186/237 | 84/108 | 232/324 | 97/172 | 23/34 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v4.0) (N=396) | Pooled Placebo (0.5 mL or 1 mL) - Adults (v4.0) (N=412) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Adults (v4.0) (N=395) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Adults (v4.0) (N=197) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v4.0) (N=403) | Pooled Placebo (0.5 mL or 1 mL) - Children (v4.0) (N=389) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Children (v4.0) (N=407) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Children (v4.0) (N=202) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v3.0) (N=187) | Pooled Placebo (0.5 mL or 1 mL) - Adults (v3.0) (N=199) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Adults (v3.0) (N=177) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Adults (v3.0) (N=99) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v3.0) (N=227) | Pooled Placebo (0.5 mL or 1 mL) - Children (v3.0) (N=214) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0) (N=237) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Children (v3.0) (N=108) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v2.0) (N=324) | Placebo (0.5 mL) - Adults (v2.0) (N=172) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v2.0) (N=34) | Placebo (0.5 mL) - Children (v2.0) (N=7)
test (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION INCOMPLETE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS INCOMPLETE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA; MALARIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS; VAGINAL DISCHARGE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLINDNESS UNILATERAL (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BURNS FIRST DEGREE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMPARTMENT SYNDROME; HUMERUS FRACTURE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS; URINARY TRACT INFECTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DROWNING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FRACTURE; TIBIA FRACTURE; FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENITAL HAEMORRHAGE; UTERINE CONTRACTIONS DURING PREGNANCY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAD INJURY; JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIV INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION; DIABETES MELLITUS INADEQUATE CONTROL; KETOACIDOSIS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA; INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Bilateral inguinal hernia and Scrotal hernia (LLT)
INGUINAL HERNIA, OBSTRUCTIVE; INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY; WOUND SECRETION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALARIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALARIA; ACUTE ABDOMEN; ANAEMIA OF PREGNANCY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALARIA; GENITAL INFECTION; APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS; GASTRIC PERFORATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PREMATURE SEPARATION OF PLACENTA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE; ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALMONELLOSIS; SALPINGITIS; PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SNAKE BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBILEUS; MALNUTRITION; FURUNCLE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TYPHOID FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE CONTRACTIONS DURING PREGNANCY; ABDOMINAL PAIN; PELVIC PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENOM POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v4.0) (N=396) | Pooled Placebo (0.5 mL or 1 mL) - Adults (v4.0) (N=412) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Adults (v4.0) (N=395) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Adults (v4.0) (N=197) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v4.0) (N=403) | Pooled Placebo (0.5 mL or 1 mL) - Children (v4.0) (N=389) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + Placebo Boost - Children (v4.0) (N=407) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine + rVSV Boost - Children (v4.0) (N=202) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v3.0) (N=187) | Pooled Placebo (0.5 mL or 1 mL) - Adults (v3.0) (N=199) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Adults (v3.0) (N=177) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Adults (v3.0) (N=99) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v3.0) (N=227) | Pooled Placebo (0.5 mL or 1 mL) - Children (v3.0) (N=214) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + Placebo Boost - Children (v3.0) (N=237) | rVSVΔG-ZEBOV-GP (rVSV) Vaccine (Diluted) + rVSV Boost (Diluted) - Children (v3.0) (N=108) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Adults (v2.0) (N=324) | Placebo (0.5 mL) - Adults (v2.0) (N=172) | Ad26.ZEBOV (rHAd26) Vaccine + MVA-BN-Filo (MVA) Boost - Children (v2.0) (N=34) | Placebo (0.5 mL) - Children (v2.0) (N=7)
Abdominal pain (Gastrointestinal disorders) | 70 (88) | 77 (99) | 80 (107) | 39 (52) | 92 (169) | 69 (127) | 97 (184) | 44 (95) | 41 (57) | 36 (49) | 38 (47) | 17 (27) | 53 (90) | 48 (88) | 56 (102) | 24 (35) | 43 (60) | 23 (30) | 7 (9) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 79 (109) | 63 (82) | 94 (128) | 45 (64) | 28 (41) | 18 (29) | 38 (61) | 14 (21) | 52 (78) | 48 (70) | 57 (84) | 29 (42) | 24 (32) | 15 (19) | 31 (51) | 12 (21) | 66 (99) | 22 (31) | 4 (10) | 0 (0)
Chills (General disorders) | 51 (55) | 48 (57) | 81 (97) | 37 (42) | 72 (114) | 59 (85) | 80 (128) | 34 (48) | 21 (24) | 21 (25) | 31 (40) | 14 (17) | 37 (50) | 21 (32) | 36 (52) | 12 (17) | 40 (45) | 16 (17) | 3 (3) | 2 (3)
Crying (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 26/137 (39) | 15/136 (28) | 27/123 (48) | 14/71 (26) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1/25 (5) | 1/24 (1) | 5/24 (5) | 1/9 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Only potentially non-verbal children less than 5 years of age assessed.
Decreased appetite (Metabolism and nutrition disorders) | 55 (69) | 54 (61) | 77 (98) | 32 (41) | 94 (162) | 80 (127) | 120 (220) | 59 (118) | 37 (58) | 39 (55) | 53 (73) | 24 (29) | 52 (82) | 31 (48) | 58 (110) | 26 (41) | 47 (58) | 21 (27) | 6 (12) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 19 (20) | 19 (21) | 7 (11) | 22 (40) | 40 (56) | 30 (39) | 21 (28) | 11 (11) | 9 (12) | 8 (8) | 3 (4) | 8 (12) | 18 (25) | 17 (22) | 5 (7) | 9 (12) | 5 (6) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 44 (53) | 46 (52) | 60 (67) | 15 (18) | 38 (70) | 27 (49) | 55 (96) | 19 (33) | 26 (35) | 35 (49) | 33 (45) | 16 (22) | 9 (15) | 17 (22) | 21 (29) | 9 (16) | 38 (45) | 17 (22) | 2 (3) | 2 (3)
Fatigue (General disorders) | 91 (119) | 84 (106) | 113 (151) | 61 (86) | 82 (131) | 66 (110) | 111 (186) | 44 (73) | 67 (107) | 69 (100) | 74 (106) | 37 (57) | 55 (96) | 25 (34) | 60 (100) | 31 (55) | 68 (115) | 39 (57) | 5 (9) | 2 (5)
Headache (Nervous system disorders) | 215 (376) | 218 (398) | 250 (447) | 116 (203) | 169 (438) | 150 (375) | 217 (555) | 97 (245) | 110 (212) | 114 (209) | 114 (214) | 66 (116) | 103 (220) | 93 (173) | 124 (264) | 56 (138) | 163 (264) | 71 (115) | 17 (30) | 2 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6) | 7 (9) | 6 (7) | 13 (22) | 11 (15) | 15 (22) | 3 (3) | 4 (4) | 5 (5) | 8 (8) | 2 (2) | 4 (6) | 5 (5) | 9 (12) | 5 (6) | 11 (12) | 7 (11) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 4 (4) | 7 (8) | 12 (14) | 3 (3) | 7 (15) | 10 (13) | 7 (11) | 9 (21) | 8 (8) | 11 (11) | 7 (7) | 6 (7) | 5 (6) | 9 (11) | 10 (13) | 3 (8) | 11 (11) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 105 (142) | 92 (115) | 138 (188) | 68 (92) | 62 (93) | 38 (46) | 78 (112) | 32 (51) | 56 (79) | 54 (72) | 61 (79) | 33 (40) | 34 (42) | 24 (28) | 50 (68) | 25 (36) | 76 (86) | 23 (24) | 6 (11) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (31) | 37 (46) | 51 (61) | 22 (29) | 26 (42) | 26 (37) | 39 (61) | 11 (15) | 19 (23) | 16 (20) | 19 (26) | 11 (14) | 19 (26) | 11 (17) | 13 (16) | 10 (15) | 19 (23) | 18 (24) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 156 (204) | 135 (188) | 180 (241) | 87 (130) | 261 (534) | 192 (399) | 278 (620) | 145 (314) | 55 (79) | 52 (82) | 69 (97) | 34 (43) | 88 (161) | 68 (101) | 114 (207) | 45 (84) | 66 (79) | 24 (27) | 8 (11) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 18 (22) | 17 (23) | 18 (21) | 9 (10) | 40 (60) | 41 (64) | 37 (58) | 15 (26) | 23 (25) | 14 (22) | 21 (27) | 6 (6) | 24 (40) | 18 (25) | 23 (33) | 12 (18) | 17 (20) | 10 (11) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (16) | 16 (16) | 25 (28) | 12 (13) | 52 (70) | 39 (53) | 55 (77) | 24 (38) | 1 (1) | 9 (11) | 6 (6) | 2 (2) | 20 (27) | 15 (21) | 19 (29) | 12 (14) | 2 (2) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-03-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02876328/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02876328/SAP_002.pdf
  • Informed Consent Form (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02876328/ICF_003.pdf